CLINICAL TRIAL: NCT06318156
Title: Exploring the Distribution Patterns and Infrared Characteristics of Force-sensitive Acupoints in Different Lumbar Nerve Segments in Patients With Lumbar Disc Herniation Based on "Press Quickly" Theory
Brief Title: Exploring the Distribution Patterns and Infrared Characteristics of Force-sensitive Acupoints in Different Lumbar Nerve Segments in Patients With LDH Based on "Press Quickly" Theory
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhou Xingchen (Other)
Responsible Party: Sponsor-Investigator, Zhou Xingchen, Prof., The Third Affiliated hospital of Zhejiang Chinese Medical University
Organization: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: ZSLL-KY-2024-056-03
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumbar Disc Herniation; Press quickly; Point-press method; Pressure-sensitive acupoints; Infrared thermal imaging
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group1(lumbar disc herniation) (Experimental): A well-trained physician donned the Finger TPS tactile pressure measurement system (Finger TPS II, BTLETG03, USA), methodically applying a consistent 60N force with a single thumb vertically downward on the acupoints of the L1 to L5 spinal segments, in accordance with the human cutaneous nerve segment map. Additionally, environmental conditions were meticulously controlled-temperature maintained between 20°C to 25°C, relative humidity at 50% to 60%, with gentle indoor lighting, quiet, and stable airflow. The MESH T-1000 Smart medical infrared thermograph, produced by Wuhan Gewu Optoelectronics Technology Co., Ltd., was utilized to assess the surface temperature of the patient's pressure-sensitive acupoint areas.
  Interventions: Diagnostic Test: Infrared thermal imaging
- Group2 (healthy control) (Experimental): A well-trained physician donned the Finger TPS tactile pressure measurement system (Finger TPS II, BTLETG03, USA), methodically applying a consistent 60N force with a single thumb vertically downward on the acupoints of the L1 to L5 spinal segments, in accordance with the human cutaneous nerve segment map. Additionally, environmental conditions were meticulously controlled-temperature maintained between 20°C to 25°C, relative humidity at 50% to 60%, with gentle indoor lighting, quiet, and stable airflow. The MESH T-1000 Smart medical infrared thermograph, produced by Wuhan Gewu Optoelectronics Technology Co., Ltd., was utilized to assess the surface temperature of the patient's pressure-sensitive acupoint areas.
  Interventions: Diagnostic Test: Infrared thermal imaging

INTERVENTIONS:
Diagnostic Test: Infrared thermal imaging — A well-trained physician donned the Finger TPS tactile pressure measurement system (Finger TPS II, BTLETG03, USA), methodically applying a consistent 60N force with a single thumb vertically downward on the acupoints of the L1 to L5 spinal segments, in accordance with the human cutaneous nerve segment map. Additionally, environmental conditions were meticulously controlled-temperature maintained between 20°C to 25°C, relative humidity at 50% to 60%, with gentle indoor lighting, quiet, and stable airflow. The MESH T-1000 Smart medical infrared thermograph, produced by Wuhan Gewu Optoelectronics Technology Co., Ltd., was utilized to assess the surface temperature of the patient's pressure-sensitive acupoint areas.

SUMMARY:
Utilizing the "responsive acupoint palpation" technique and infrared thermography, we investigated the distribution patterns of pressure-sensitive acupoints across different lumbar spinal segments in patients with lumbar disc herniation (LDH). Methodology: The Finger TPS tactile pressure measurement system was employed to conduct sensitivity examinations on the acupoints of the L1~L5 lumbar spine in 80 LDH patients (Group 1) and 80 healthy individuals (Group 2), applying a standardized force of 60N. When a sensation of comfort was elicited, the points were marked on a human cutaneous nerve segment map. We then utilized infrared thermography to collect and compare the temperature differences of the top 10 most frequently responsive acupoint areas in the experimental group against those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18 to 65 years, regardless of gender.
* Radiological confirmation of central type L4~L5 intervertebral disc herniation.
* Meeting the diagnostic criteria for lumbar disc herniation, primarily manifesting as lower back pain, radicular pain, and numbness or weakness in the lower limbs, with imaging findings consistent with neurological localization.
* Patients in the non-acute phase of mild to moderate pain and functional impairment (onset more than 2 weeks ago), with a visual analog scale (VAS) score greater than 4 points and a Japanese Orthopaedic Association (JOA) score less than 15 points.
* No consumption of analgesics, neurotrophic drugs, or sedatives, and no systemic treatment in the past week.
* Willing participants in the study who have signed an informed consent form.

Exclusion Criteria:

* Concomitant internist and gynecological diseases that can cause lower back pain, such as nephritis, urinary tract stones, gynecological inflammations, and uterine pathologies.
* Individuals with severe primary diseases of the cardiovascular, cerebrovascular, liver, kidney, etc.
* Patients with neurosis or psychiatric disorders, or those with a history of cranial trauma or coma.
* Patients with primary or ankylosing sciatica.
* Individuals with concomitant lumbar spondylolisthesis.
* Patients with lumbar spine tumors or tuberculosis.
* Individuals with consciousness disorders, severe impairments in vision, hearing, or speech, or any other condition that prevents the completion of a health assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
skin temperature | up to one month
  The medical infrared thermographic camera captures thermal images of the human cutaneous nerve segment map on the back of the subjects, focusing on the L1 to L5 spinal segment areas.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jiang Lv, Ph.D., Study Chair — The Third Clinical Medical College of Zhejiang Chinese Medical University, Hangzhou, Zhejiang,China
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No